CLINICAL TRIAL: NCT06056947
Title: Phase III Study to Evaluate Efficacy and Safety of Different Formulations of Fenticonazole + Tinidazole + Lidocaine in the Treatment of Bacterial Vaginosis, Candidal Vulvovaginitis, Trichomonal Vaginitis and Mixed Infections
Brief Title: Evaluation of Efficacy and Safety of Two New Formulations Compared to Gynomax® XL Ovule
Acronym: One-Shot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Monitor CRO (Industry); Exeltis Turkey (Industry)
Responsible Party: Principal Investigator, Erol Tavmergen, MD, MD Prof, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MON580.130.3
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Trichomonal Vaginitis; Bacterial Vaginosis; Candidal Vulvovaginitis; Mixed Vaginal Infections
MeSH Terms: conditions — Trichomonas Vaginitis; Vaginosis, Bacterial; Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fenticonazole + tinidazole + lidocaine vaginal ovule (EVEGYN A) (Experimental): EVEGYN A is a fixed-dose combination of 600 mg fenticonazole nitrate + 1000 mg tinidazole + 100 mg lidocaine vaginal ovule.
  Interventions: Drug: EVEGYN A
- fenticonazole + tinidazole + lidocaine vaginal ovule (EVEGYN B) (Experimental): EVEGYN B is a fixed-dose combination of 600 mg fenticonazole nitrate + 2000 mg tinidazole + 100 mg lidocaine vaginal ovule.
  Interventions: Drug: EVEGYN B
- Gynomax® XL Vaginal Ovule (Active Comparator): Gynomax® XL is a fixed-dose combination of 300 mg tinidazole + 200 mg tioconazole nitrate + 100 mg lidocaine
  Interventions: Drug: Gynomax® XL Vaginal Ovule

INTERVENTIONS:
Drug: EVEGYN A — EVEGYN A: Fixed-dose combination of 600 mg fenticonazole nitrate + 1000 mg tinidazole + 100 mg lidocaine vaginal ovule Single dose, single administration (1x1)
  Arms: fenticonazole + tinidazole + lidocaine vaginal ovule (EVEGYN A)
Drug: EVEGYN B — EVEGYN B: Fixed-dose combination of 600 mg fenticonazole nitrate + 2000 mg tinidazole + 100 mg lidocaine vaginal ovule Single dose, single administration (1x1)
  Arms: fenticonazole + tinidazole + lidocaine vaginal ovule (EVEGYN B)
Drug: Gynomax® XL Vaginal Ovule — 200 mg tioconazole + 300 mg tinidazole + 100 mg lidocaine single dose / day, during three consecutive days (1x1 / 3 days)
  Arms: Gynomax® XL Vaginal Ovule

SUMMARY:
Efficacy and safety of two new formulations compared to Gynomax® XL ovule in the treatment of trichomonal vaginitis, bacterial vaginosis, candidal vulvovaginitis and mixed vaginal infections was evaluated in this randomized, three-arms, multicentral study.

DETAILED DESCRIPTION:
This was a national, randomized, 3-arms, phase III study conducted in 16 centers in Türkiye.

It was aimed to evaluate the efficacy and safety of different fixed dose vaginal ovule formulations of fenticonazole + tinidazole + lidocaine (Formulation A and Formulation B) in the treatment of bacterial vaginosis, candidal vulvovaginitis, trichomonal vaginitis and mixed infections with comparison to Gynomax® XL vaginal ovule.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with age of ≥ 18 and ≤ 55 years who have a regular menstrual cycle (at least 10 times a year)
2. Female patients who previously experienced vaginal intercourse
3. Patients requiring treatment for bacterial vaginosis, candidal vulvovaginitis, trichomonal vaginitis or mixed infections according to the investigator's decision
4. Signed informed consent

Exclusion Criteria:

1. Known hypersensitivity to active ingredients (including their derivatives) of the study medications
2. Vaginismus, endometriosis, dyspareunia
3. Detection of urinary tract infection in urinalysis
4. Pancreatitis, hypertriglyceridemia, liver diseases, benign or malign tumors and ongoing organ failure
5. Usage of herbal medicines and drugs that interfere with microsomal enzymes, especially cytochrome P450 (phenytoin, phenobarbital, primidone, carbamazepine, rifampicin, topiramate, felbamate, griseofulvin, HIV protease inhibitors such as ritonavir, nucleoside reverse transcriptase inhibitors such as efavirenz)
6. History of cardiovascular event
7. Uncontrolled diabetes and hypertension
8. Presence or known risk or of venous or arterial thromboembolism
9. Undiagnosed abnormal vaginal bleeding, bleeding disorders, bleeding due to intrauterine device implantation during study period, presence of genital tumors
10. Use of drugs containing ombitasvir / paritaprevir / ritonavir or dasabuvir during or two weeks before initiation of the study
11. Pregnancy and/or breastfeeding
12. Participation in any other trial 30 days before initiation of the study
13. Postmenopausal women
14. Chronic alcoholism
15. Patients with organic neurological disorders
16. Patients with blood dyscrasia or with a history of blood dyscrasia
17. Usage of medications containing acenocoumarol, anisindione, dicoumarol, phenindione, phenprocoumon, warfarin, cholestyramine, cimetidine, cyclosporine, disulfiram, fluorouracil, fosphenitoin, ketoconazole, lithium, rifampin, tacrolimus or propranolol
18. Presence of a sexually transmitted disease such as syphilis, gonorrhea, chlamydia etc. according to the investigator's decision
19. Patients who cannot perform sexual abstinence during the study
20. Patients whose treatment may be affected due to sagging of uterus or any other anatomical disorder

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 577 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who had complete response to treatment according to clinical findings | 13 days (+/- 5 days) after treatment
  Efficacy

SECONDARY OUTCOMES:
Percentage of patients who had partial response to treatment according to clinical findings | 13 days (+/- 5 days) after treatment
  Efficacy
Percentage of patients who recovered according to microbiological findings | 13 days (+/- 5 days) after treatment
  Efficacy
Frequency and percentage of patients with SAEs/AEs in each arm | 13 days (+/- 5 days)
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Family Planning and Infertility Application and Research Center, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No